CLINICAL TRIAL: NCT04937140
Title: 14-3-3 η (Eta) Protein as a Marker of Disease Activity, Severity and Subclinical Atherosclerosis in Patients With Rheumatoid Arthritis.
Brief Title: Assessment of 14-3-3 η (Eta) Protein Antibodies in the Serum of Rheumatoid Arthritis Patients and Its Relation to Atherosclerosis.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Doaa Adel Ibrahim, Specialist of Rheumatology & Rehabilitation In the Medical Administration Sohag Universit, Sohag University
Other Study IDs: Soh-Med-21-06-11
Record Dates: First submitted 2021-06-14; First posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Rheumatoid Arthritis
Keywords: RA
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- rheumatoid arthritis patients: 90 RA patients diagnosed according to the American college of rheumatology (ACR) -EULAR RA classification criteria 2010
  Interventions: Diagnostic Test: 14-3-3 η (eta) protein antibodies in the serum of rheumatoid arthritis patients
- control group: 50 age and sex matched healthy controls. All
  Interventions: Diagnostic Test: 14-3-3 η (eta) protein antibodies in the serum of rheumatoid arthritis patients

INTERVENTIONS:
Diagnostic Test: 14-3-3 η (eta) protein antibodies in the serum of rheumatoid arthritis patients — assessment of 14-3-3 η (eta) protein antibodies in the serum of rheumatoid arthritis patients and Carotid Doppler ultrasound (for measurement of carotid intima media thickness and detection of plaques)
  Other Names: Carotid Doppler ultrasound (for measurement of carotid intima media thickness and detection of plaques)

SUMMARY:
The aims of this study are: • To assess 14-3-3 η (eta) protein antibodies in the serum of rheumatoid arthritis patients and its relation to disease activity and severity. • To investigate the role of 14-3-3 η (eta) protein in the diagnosis or assessment of subclinical carotid artery atherosclerosis.

DETAILED DESCRIPTION:
All the patients will be interviewed for demographic and clinical data (age, sex, occupation, age at onset of the disease, joints affected, extra-articular features, disease duration, family history and treatment regimen). • Assessment of medical and rheumatologic history.

* Careful general and musculoskeletal examination.
* Assessment of disease activity will be performed using the Disease Activity Score (DAS28) including 28 tender and swollen joint count, ESR and visual analogue scale.
* X-ray both hands and feet
* Larsen Score
* Assessment of Body Mass Index (BMI)
* Laboratory investigations:
* Complete blood count (CBC) • Rheumatoid factor (RF) by latex method • Anti citrullinated protein antibodies ACPA by enzyme-linked immunosorbent assay (ELISA) • 14-3-3 η (eta) protein by (ELISA) • Erythrocytic sedimentation rate (ESR) • Quantitative C-reactive protein (CRP) • fasting blood glucose • lipid profile • Carotid Doppler ultrasound (for measurement of carotid intima media thickness and detection of plaques) • ECG

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:

  1. Patients with RA classified according to the revised American College of Rheumatology (ACR)/EULAR RA classification criteria 2010 for RA.
  2. Age ≥ 18 years.
  3. Patients who are able and willing to give written informed consent.
  4. Disease duration more than one year

     Exclusion Criteria:

  <!-- -->

  1. Any other autoimmune disease rather than RA.
  2. Patients with any disease affecting the cardiovascular system other than RA.
  3. Patients with known risk factors for atherosclerosis as diabetes, hypertension, hyperlipidemia and obesity.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study will include 90 RA patients diagnosed according to the American college of rheumatology (ACR) -EULAR RA classification criteria 2010 in addition to 50 age and sex matched healthy controls.
  All the patients will be recruited from Rheumatology and Rehabilitation outpatient clinic in Sohag University Hospitals, Faculty of Medicine .
  Patients
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
14-3-3 eta protein as measured by enzyme-linked immunosorbent assay (ELISA) in the serum of the participants and carotid intima media thickness as determined by carotid doppler ultrasound | through study completion, an average of 1 year"
  relation between presence of 14-3-3 η (eta)by enzyme-linked immunosorbent assay (ELISA) in the serum of the participants and carotid intima media thickness and detection of plaques

CONTACTS AND LOCATIONS:
Overall Officials: doaa adel, specialist, Principal Investigator — In the Medical Administration Sohag University

IPD SHARING:
Plan to Share IPD: No